CLINICAL TRIAL: NCT03203148
Title: Comparison of Two Point of Care Techniques Mechanical Versus Biochemical Activated Clotting Time
Brief Title: Two Monitors for Measuring the Activated Clotting Time: A Comparison
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-HeartCentre-003
Record Dates: First submitted 2017-06-13; First posted 2017-06-29 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Cardiopulmonary Bypass; Blood Coagulation; Point-of-Care Testing
Keywords: Cardiopulmonary Bypass; Blood Coagulation Testing; Point-of-Care Testing
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABG Surgical Patients: Patients undergoing coronary bypass grafting with cardiopulmonary bypass
  Interventions: Diagnostic Test: Point-of-Care ACT

INTERVENTIONS:
Diagnostic Test: Point-of-Care ACT — Comparison between two point-of-care devices for measurement of the activated clotting time

SUMMARY:
In this observational study a comparison is made between two different monitors for measurement of the activated clotting time (ACT): mechanical versus biochemical techniques

DETAILED DESCRIPTION:
The ACT is a functional test influenced by multiple factors, such as platelet function, coagulation factors, temperature and contact activation inhibitors. Results produced by different monitors are also prone to vary influenced by the specific method employed to perform the test.

The present clinical study aims to compare two types of ACT monitors: the Hemostatic Management System Plus (Medtronic) and i-STAT (Abbott) in 20 cardiac surgical patients by performing five intraoperative consecutive measurements using anti factor Xa as a reference for the actual heparin concentration.

Inclusion criteria comprised patients aged 20-80 years, scheduled for coronary bypass surgery.

Measurements: 1) before induction of anaesthesia 2 ) after heparin bolus 3) rewarming of the patient 4) weaning from cardiopulmonary bypass 5) after protamine administration.

The Hemostatic System Plus ACT monitor served as reference for dosing of heparin in all patients. The study protocol did not intervene with the standard protocol used for anticoagulation. No patient interventions were made.

It is hypothesised that the i-STAT ACT monitor has a better correlation with the actual heparin concentration than the Hemostatic Management System Plus

ELIGIBILITY:
Inclusion Criteria: Patients listed for coronary bypass surgery, -

Exclusion Criteria: Primary coagulation disorder, diabetes mellitus, ongoing anti-coagulation therapy, emergency, reduced kidney function, allergy for fish, sea food and protamine

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for routine coronary bypass surgery with the use of cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Activated Clotting time | Intraoperative
  Coagulation Measure

SECONDARY OUTCOMES:
Anti-Factor Xa | Intraoperative
  Reference for heparin plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Hedström, MD, Study Director — Heart Centre, Umeå University Hospital, Sweden
Locations (1):
- Heart Centre Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teufelsbauer H, Proidl S, Havel M, Vukovich T. Early activation of hemostasis during cardiopulmonary bypass: evidence for thrombin mediated hyperfibrinolysis. Thromb Haemost. 1992 Sep 7;68(3):250-2. PMID 1440486
- [Background] Hattersley PG. Progress report: the activated coagulation time of whole blood (ACT). Am J Clin Pathol. 1976 Nov;66(5):899-904. doi: 10.1093/ajcp/66.5.899. PMID 983997
- [Background] Guzzetta NA, Monitz HG, Fernandez JD, Fazlollah TM, Knezevic A, Miller BE. Correlations between activated clotting time values and heparin concentration measurements in young infants undergoing cardiopulmonary bypass. Anesth Analg. 2010 Jul;111(1):173-9. doi: 10.1213/ANE.0b013e3181e13470. Epub 2010 Jun 2. PMID 20519414
- [Background] Svenmarker S, Appelblad M, Jansson E, Haggmark S. Measurement of the activated clotting time during cardiopulmonary bypass: differences between Hemotec ACT and Hemochron Jr apparatus. Perfusion. 2004;19(5):289-94. doi: 10.1191/0267659104pf755oa. PMID 15506033
- [Background] Raymond PD, Ray MJ, Callen SN, Marsh NA. Heparin monitoring during cardiac surgery. Part 1: Validation of whole-blood heparin concentration and activated clotting time. Perfusion. 2003 Sep;18(5):269-76. doi: 10.1191/0267659103pf672oa. PMID 14604242